CLINICAL TRIAL: NCT01445106
Title: A Phase I Trial of Nelfinavir (Viracept) in Adults With Solid Tumors
Brief Title: A Phase I Trial of Nelfinavir (Viracept ) in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 070047; 07-C-0047; NCT00436735 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-12-02

CONDITIONS: Solid Tumors
Keywords: HIV Protease Inhibitor; Drug Repositioning; Akt/Mtor Inhibitor; Targeted Therapy; Off - Label Drugs; Nelfinavir; Protease Inhibitor; Solid Tumor; Phase I; Malignant Tumor
MeSH Terms: conditions — Neoplasms | interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir
Drug: Nelfinavir Mesylate

SUMMARY:
Background:

* The PI3K/Akt/mTOR pathway is an important target in cancer because it promotes chemotherapeutic resistance and confers a poor prognosis for many types of cancers.
* Several inhibitors of the pathway are being developed as cancer therapeutics. However, the process of de novo drug development takes years, and is often curtailed due to diminished activity and/or unforeseen toxicities in clinical trials.
* One approach to expedite the development of new cancer therapies is to test drugs that are already approved for other indications.
* Our group has shown that nelfinavir, an orally available FDA-approved HIV-1 protease inhibitor used to treat HIV/AIDS, can inhibit endogenous Akt and growth factor receptor induced Akt activity in cancer cells.
* Importantly, nelfinavir demonstrates dose-dependent cytotoxicity in every cell line in the NCI 60 cell line panel at plasma concentrations attainable in human plasma, is profoundly effective in cancer cell lines that have been selected to become resistant to standard therapies, and inhibits tumor growth in-vivo.

Objectives:

* Because an MTD with nelfinavir has not been observed in prior phase I studies with HIV patients, the objectives of the Phase I design will be:
* To establish the MTD and dose limiting toxicity for this drug in patients with solid Tumors.
* To correlate nelfinavir pharmacokinetics with baseline activity of CYP3A4 as assessed by measuring midazolam clearance.
* To preliminarily explore the biological and clinical effects through a series of correlative studies involving analysis of blood and tissue across patients throughout the study.

Eligibility:

-Adults with solid tumors who are refractory to, or have relapsed after receiving, standard front-line chemotherapies are eligible.

Design:

* Patients will receive nelfinavir beginning at the FDA-approved dose for HIV patients (1250 mg po bid).
* Dose escalations will occur for 6 dose levels i.e. cohorts, or until the MTD is reached.
* Up to 45 patients are expected to be enrolled.
* Staging CT scans will be performed every two cycles.

DETAILED DESCRIPTION:
Background:

-The PI3K/Akt/mTOR pathway is an important target in cancer because it promotes

chemotherapeutic resistance and confers a poor prognosis for many types of cancers.

* Several inhibitors of the pathway are being developed as cancer therapeutics. However, the process of de novo drug development takes years, and is often curtailed due to diminished activity and/or unforeseen toxicities in clinical trials.
* One approach to expedite the development of new cancer therapies is to test drugs that are already approved for other indications.
* Our group has shown that nelfinavir, an orally available FDA-approved HIV-1 protease

inhibitor used to treat HIV/AIDS, can inhibit endogenous Akt and growth factor receptor

induced Akt activity in cancer cells.

-Importantly, nelfinavir demonstrates dose-dependent cytotoxicity in every cell line in the

NCI 60 cell line panel at plasma concentrations attainable in human plasma, is profoundly

effective in cancer cell lines that have been selected to become resistant to standard therapies, and inhibits tumor growth in-vivo.

Objectives:

-Because an MTD with nelfinavir has not been observed in prior phase I studies with HIV

patients, the objectives of the Phase I design will be:

-To establish the MTD and dose limiting toxicity for this drug in patients with solid

Tumors.

-To correlate nelfinavir pharmacokinetics with baseline activity of CYP3A4 as

assessed by measuring midazolam clearance.

-To preliminarily explore the biological and clinical effects through a series of

correlative studies involving analysis of blood and tissue across patients throughout

the study.

Eligibility:

-Adults with solid tumors who are refractory to, or have relapsed after receiving, standard

front-line chemotherapies are eligible.

Design:

* Patients will receive nelfinavir beginning at the FDA-approved dose for HIV patients (1250 mg po bid).
* Dose escalations will occur for 6 dose levels i.e. cohorts, or until the MTD is reached.
* Up to 45 patients are expected to be enrolled.
* Staging CT scans will be performed every two cycles.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have a histologically confirmed solid malignancy by the Laboratory of Pathology at the Clinical Center/NIH or the Laboratory of Pathology at NNMC.

Patients must: have either relapsed following, or progressed through, standard therapy; have a current disease state for which there is no standard effective therapy; have refused standard therapy in cases where no curative option exists.

Patients may have had any number of chemotherapeutic regimens.

Age greater than or equal to 18 years of age.

ECOG performance score of less than or equal to 2.

An expected survival of greater than or equal to 3 months.

Patients must have the capacity and willingness to sign a written informed consent and demonstrate willingness to comply with an oral regimen.

Patients must have normal organ and marrow function as defined below:

* absolute neutrophil count greater than or equal to 1,500/mL.
* platelets greater than or equal to 100,000/mL.
* total bilirubin less than 1.5 X upper limit of institutional normal.
* AST(SGOT) less than or equal to 2.5 X upper limit of institutional normal.
* ALT(SGPT) less than or equal to 2.5 X upper limit of institutional normal.
* Creatinine less than 1.5 X upper limit of institutional normal.

Patients must agree to use non-hormonal methods of birth control, e.g., barrier methods, for the duration of the study due to possible drug interactions.

Patients will be asked if they would consent to a biopsy before and after treatment in order to provide biologic correlates for analysis, but these will be optional, and the patients will be eligible whether they consent to do this or not.

Patients with brain metastasis must have undergone evaluation and appropriate counseling and treatment by radiation oncology.

EXCLUSION CRITERIA:

Pregnant or lactating women.

Patients who have had chemotherapy or biologic agents in the last 28 days prior to entering the study.

Any concurrent therapy with chemotherapeutic agents or biologic agents or radiation therapy.

Patients with a myocardial infarction in the six months prior to enrollment.

Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Patients that are on the following CYP3A4 inhibitors and cannot replace these medications with other equivalent medications for the period of the study: antiarrhythmics (amiodarone, quinidine), neuroleptics (pimozide), sedative/hypnotic agents (midazolam, triazolam), ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine), HMG-CoA reductase inhibitors (lovastatin, simvastatin, atorvastatin), rifampin, rifabutin, felodipine, nifedipine, and sildenafil or St. John's wort. Patients whose baseline medication regimen includes 2 or more medications of a class carries the potential for serious side effects, and which must be changed becaused of potential interaction with nelfinavir, they must be stable on the new regimen for 7 days before enrollment.

Patients that are on escalating doses of corticosteroids for other non-cancerous medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-12-11; Primary Completion 2011-05-09 (Actual); Study Completion 2011-05-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety and toxicity of nelfinavir in human subjects with solid tumors and to determine the maximum tolerated dose in this group of patients.

SECONDARY OUTCOMES:
To determine the PK of nelfinavir admin, correlate cytochrome P450 3A4 activity with nelfinavir levels and establish prelim evidence of clinical efficacy of this regimen in solid tumor malignancy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Balsara BR, Pei J, Mitsuuchi Y, Page R, Klein-Szanto A, Wang H, Unger M, Testa JR. Frequent activation of AKT in non-small cell lung carcinomas and preneoplastic bronchial lesions. Carcinogenesis. 2004 Nov;25(11):2053-9. doi: 10.1093/carcin/bgh226. Epub 2004 Jul 7. PMID 15240509
- [Background] Bernal-Mizrachi E, Fatrai S, Johnson JD, Ohsugi M, Otani K, Han Z, Polonsky KS, Permutt MA. Defective insulin secretion and increased susceptibility to experimental diabetes are induced by reduced Akt activity in pancreatic islet beta cells. J Clin Invest. 2004 Oct;114(7):928-36. doi: 10.1172/JCI20016. PMID 15467831
- [Background] Bernal-Mizrachi E, Wen W, Stahlhut S, Welling CM, Permutt MA. Islet beta cell expression of constitutively active Akt1/PKB alpha induces striking hypertrophy, hyperplasia, and hyperinsulinemia. J Clin Invest. 2001 Dec;108(11):1631-8. doi: 10.1172/JCI13785. PMID 11733558